CLINICAL TRIAL: NCT05490667
Title: The Efficacy and Safety of Anlotinib Combined With Chemotherapy in the Treatment of Unresectable Advanced Desmoid Tumors: a Prospective Single-arm Clinical Study
Brief Title: Clinical Study of Anlotinib Combined With Chemotherapy in the Treatment of Unresectable Advanced Desmoid Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhang Peng, Associate chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-STS-002
Record Dates: First submitted 2022-08-02; First posted 2022-08-08 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-08

CONDITIONS: Desmoid
MeSH Terms: conditions — Desmoid Tumors | interventions — anlotinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Anlotinib combined with chemotherapy for desmoid tumors
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib combined with chemotherapy for desmoid tumors
  Other Names: chemotherapy

SUMMARY:
Thirty patients with desmoid tumors (invasive fibromatosis) will be recruited in the Department of Bone and Soft Tissue, Henan Cancer Hospital. This is a prospective, multicenter, single-arm clinical study to evaluate the efficacy and safety of anlotinib combined with chemotherapy in the treatment of inoperable advanced desmoid tumors.

DETAILED DESCRIPTION:
Thirty patients with desmoid tumor (invasive fibromatosis) will be recruited in the Department of Bone and Soft Tissue, Henan Cancer Hospital. This is a prospective, multicenter, single-arm clinical study to evaluate the efficacy and safety of anlotinib combined with chemotherapy in the treatment of inoperative advanced desmoid tumor. To evaluate the 6-month progression-free survival rate, 12-month progression-free survival rate, progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR) and safety of anlotinib combined with chemotherapy for desmoid tumors.

ELIGIBILITY:
Inclusion Criteria:

Advanced desmoid tumor confirmed by pathology.

The presence of measurable lesions meeting RECIST 1.1 criteria.

Male and female, aged ≥10 years.

Eastern Cooperative Oncology Group(ECOG) physical condition 0-2 points.

Radiographic evidence of recurrence or disease progression within the past 6 months (according to RECIST criteria).

Imaging evaluation met the inoperable criteria as follows:

Radical surgery will cause large defects of skin, muscle and other soft tissues, resulting in great changes in limb appearance and loss of function, or require major reconstructive surgery such as patch repair and flap repair; Radical surgery will involve the main blood vessels and nerves; The tumor involves the bone, and the safe margin cannot be achieved under the premise of bone preservation; By explaining the condition to the patient, the patient refuses to try the operation after weighing the advantages and disadvantages; Amputation is not considered.

Major organ function is normal, that is, meet the following criteria: hemoglobin (Hb) ≥ 95g/L,

Neutrophil (ANC) ≥1.5×109/L, platelet count (PLT) ≥ 80×109/L,

Serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN), blood urea nitrogen (BUN) ≤ 2.5× upper limit of normal(ULN);

Total bilirubin (TB) ≤ ULN;

Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; Albumin (ALB) ≥ 35g/L

Prothrombin time (PT) and partial prothrombin time (PTT) ≤1.2×ULN left ventricular ejection fraction ≥50%;

Patients gave informed consent and signed a written consent form.

Patients had good compliance and voluntarily accepted follow-up, treatment, laboratory tests, and other research steps as planned.

Exclusion Criteria:

Patients who have used anlotinib, pesopanib, sorafenib, sunitinib, apatinib and other TKI drugs in the past;

with pleural effusion or ascites, causing respiratory syndrome (≥CTCAE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath with little activity; affects instrumental activities of daily living]);

The presence or current presence of other malignant tumors within 3 or 5 years, with the exception of cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors (Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading basement membrane));

Systemic antitumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy, was planned within 4 weeks before enrollment or during the study medication period (or silk was used within 6 weeks before treatment with the trial drug) Schizomycin C). Overextended field radiotherapy (EF-RT) was performed within 4 weeks before grouping or field-limited radiotherapy to evaluate tumor lesions was performed within 2 weeks before enrollment.

Unrelieved toxic reactions above CTCAE(4.0) grade 1 due to any previous treatment, excluding alopecia;

with multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);

Patients with any severe and/or uncontrolled disease, including:

Patients with poor blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg);

Patients with grade I or higher myocardial ischemia or infarction, arrhythmias (including QTC ≥480ms), or congestive heart failure grade 2 (New York Heart Association (NYHA) classification);

Active or uncontrolled severe infection (≥CTCAE grade 2 infection);

Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need antiviral therapy;

Renal failure requiring hemodialysis or peritoneal dialysis;

Have a history of immunodeficiency, including being HIV positive or suffering from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;

poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);

The urine routine indicated urinary protein ≥++, and confirmed 24-hour urinary protein quantity > 1.0 g;

patients with epileptic seizures requiring treatment;

Patients with hypothyroidism: Thyroid stimulating hormone（TSH）>4.2mlU/L;

Subjects with any medical condition that may increase the risk of gastrointestinal bleeding or perforation: such as active gastrointestinal ulcers, known luminal metastatic lesions, inflammatory bowel disease, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days before the study;

Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.);

Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days before enrollment;

Patients whose imaging showed that the tumor had invaded the periphery of important blood vessels or who were judged by the investigator to be very likely to invade important blood vessels during the subsequent study and cause fatal massive bleeding;

Patients with any evidence of bleeding constitution or history, regardless of severity; Four weeks before grouping In patients with any bleeding or bleeding events ≥CTCAE grade 3, unhealed wounds, ulcers, or fractures; Significant blood coughing or daily hemoptysis of 2.5ml or more within 2 months before enrollment;

Experienced an arteriovenous thrombotic event within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;

Abnormal coagulation (INR > 1.5 or PT >1.2 ULN or PTT >1.2 ULN), bleeding tendency or undergoing thrombolytic or anticoagulant therapy;

Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or similar agents;

Those who had received a potent CYP3A4 inhibitor within 7 days or received a potent CYP3A4 inducer within 12 days prior to study enrollment. Drugs with CYP3A4, CYP2D6, or CYP2C8 substrates should be avoided;

Use drugs that may lead to prolongation of QT interval and tip torsion in ECG within 4 weeks;

Those who have a history of psychotropic drug abuse and are unable to quit or have mental disorders;

Participated in clinical trials of other antitumor drugs within four weeks;

Pregnant or lactating patients;

Any condition that, in the investigator's judgment, may impair the subject's ability to meet or perform the study requirements.

Ages: 10 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 24months
  From initiation of treatment to tumor progression

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Bone and Soft Tissue ,Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No